CLINICAL TRIAL: NCT05850637
Title: Phase II Study to Evaluate the Effectiveness and Toxicity of Adjuvant Ultra-hypofractionated Radiotherapy for the Treatment of Early and Locally Advanced Breast Cancer
Brief Title: Evaluate the Effectiveness and Toxicity of Adjuvant Ultra-hypofractionated Radiotherapy for Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prevent Senior Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INSTITUTO PREVENT SENIOR - IPS
Record Dates: First submitted 2023-04-20; First posted 2023-05-09 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer Female
Keywords: Breast Cancer; Adjuvant radiotherapy; Ultra-hypofractionated
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective phase 2 non-randomized single-arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm Ultra-hypofractionated (Experimental): 5 fractions of 5.7 Gy every other day in the breast or chest wall region, with or without the inclusion of regional lymph node drainage chains
  Interventions: Radiation: adjuvant ultra-hypofractionated radiotherapy

INTERVENTIONS:
Radiation: adjuvant ultra-hypofractionated radiotherapy — adjuvant ultra-hypofractionated radiotherapy for the treatment of early and locally advanced breast cancer

SUMMARY:
Prospective phase 2 study to evaluate the safety and efficacy of ultra-hypofractionated adjuvant radiotherapy in 5 fractions of 5.7 Gy in patients aged over 65 years.

DETAILED DESCRIPTION:
Prospective phase 2 non-randomized single-arm study to evaluate the safety and efficacy of ultra-hypofractionated adjuvant radiotherapy in 5 fractions of 5.7 Gy in patients aged over 65 years.

ELIGIBILITY:
Inclusion Criteria:

1. Female patient;
2. Pathological confirmation of invasive breast carcinoma regardless of histological subtype and hormonal profile;
3. Age greater than or equal to 65 years;
4. Breast-conserving surgery or mastectomy with or without axillary approach
5. With or without neoadjuvant or adjuvant systemic treatment

Exclusion Criteria:

1. Patients with previous thoracic irradiation;
2. Patients with indication for bilateral thoracic irradiation;
3. Patients with breast reconstruction with prosthesis or autologous tissue;
4. Patients with compromised surgical margins after resection;
5. pT1-pT2 pN0 patients undergoing radical mastectomy.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2021-02-11 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Acute toxicity | Events of radiotherapy up to 3 months
  Acute skin toxicity was evaluated the criteria followed the Standard Common Terminology Criteria for Adverse Events - CTCAE v 5.0
Late toxicity | Events after 3 months of radiotherapy completion
  Delayed skin and subcutaneous toxicities were evaluated according to the Radiation Therapy Oncology Group (RTOG) classification.

SECONDARY OUTCOMES:
Locoregional free survival | 3 years
  from the date of initiation of treatment until the date of recurrence or progression of locoregional disease evidence
Distant free survival | 3 years
  from the date of initiation of treatment until the date of progression of distant disease evidence
Overall survival | 3 years
  defined from the date of initiation of treatment until the patient's death
Cosmesis change | week 10 and week 26 after the end of the treatment
  was assessed using the Harvard/NSABP/RTOG scale. The Harvard/NSABP/RTOG scale score is a 4-point breast cosmetic scale, which was assessed by clinicians at baseline (after surgery) and two additional times during follow-up.
  1. Excellent: When compared to the untreated breast, there is no difference or minimal difference in the size or shape of the treated breast. The breast texture is the same or slightly different. There may be thickening, scar tissue, or fluid buildup in the breast, but not enough to change the appearance.
  2. Good: There is a slight difference in the size or shape of the treated breast compared to the untreated breast or compared to the original appearance of the treated breast. There may be a slight reddening or darkening of the breast. Thickening or scar tissue inside the breast causes only a slight change in shape or size.
  3. Fair: Obvious difference in the size and shape of the treated breast. This change involves a quarter or less of the breast. There may be
QOL (Quality of Life) changes | 3 years
  was assessed using the scales proposed by the EORTC (European Organization for Research and Treatment of Cancer). The EORTC QOQ-C30 and EORTC QLQ-BR-23 scales.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.

OTHER OUTCOMES:
Breast volume and toxicity relationship | 3 years
  We analyzed the impact of CTV (Clinical Target Volume) volume (representing breast size), and dosimetric data, with a special focus on the maximum dose and dose in homogeneity (defined as the absolute volumes of breast tissue exposed to ≥100%, ≥104% and ≥107% of the prescribed dose

CONTACTS AND LOCATIONS:
Overall Officials: Marcel MF Fang, MD, Principal Investigator — Instituto de Pesquisa Prevent Senior
Locations (1):
- Instituto de Pesquisa Prevent Senior, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] START Trialists' Group; Bentzen SM, Agrawal RK, Aird EG, Barrett JM, Barrett-Lee PJ, Bentzen SM, Bliss JM, Brown J, Dewar JA, Dobbs HJ, Haviland JS, Hoskin PJ, Hopwood P, Lawton PA, Magee BJ, Mills J, Morgan DA, Owen JR, Simmons S, Sumo G, Sydenham MA, Venables K, Yarnold JR. The UK Standardisation of Breast Radiotherapy (START) Trial B of radiotherapy hypofractionation for treatment of early breast cancer: a randomised trial. Lancet. 2008 Mar 29;371(9618):1098-107. doi: 10.1016/S0140-6736(08)60348-7. Epub 2008 Mar 19. PMID 18355913
- [Background] AMIN, M. B. et al. American Joint Committee on Cancer (AJCC). AJCC Cancer Staging Manual. [s.l: s.n.].
- [Background] Bartelink H, Maingon P, Poortmans P, Weltens C, Fourquet A, Jager J, Schinagl D, Oei B, Rodenhuis C, Horiot JC, Struikmans H, Van Limbergen E, Kirova Y, Elkhuizen P, Bongartz R, Miralbell R, Morgan D, Dubois JB, Remouchamps V, Mirimanoff RO, Collette S, Collette L; European Organisation for Research and Treatment of Cancer Radiation Oncology and Breast Cancer Groups. Whole-breast irradiation with or without a boost for patients treated with breast-conserving surgery for early breast cancer: 20-year follow-up of a randomised phase 3 trial. Lancet Oncol. 2015 Jan;16(1):47-56. doi: 10.1016/S1470-2045(14)71156-8. Epub 2014 Dec 9. PMID 25500422
- [Background] Benedict SH, Yenice KM, Followill D, Galvin JM, Hinson W, Kavanagh B, Keall P, Lovelock M, Meeks S, Papiez L, Purdie T, Sadagopan R, Schell MC, Salter B, Schlesinger DJ, Shiu AS, Solberg T, Song DY, Stieber V, Timmerman R, Tome WA, Verellen D, Wang L, Yin FF. Stereotactic body radiation therapy: the report of AAPM Task Group 101. Med Phys. 2010 Aug;37(8):4078-101. doi: 10.1118/1.3438081. PMID 20879569
- [Background] Collaborative Group on Hormonal Factors in Breast Cancer. Familial breast cancer: collaborative reanalysis of individual data from 52 epidemiological studies including 58,209 women with breast cancer and 101,986 women without the disease. Lancet. 2001 Oct 27;358(9291):1389-99. doi: 10.1016/S0140-6736(01)06524-2. PMID 11705483
- [Background] Bray F, McCarron P, Parkin DM. The changing global patterns of female breast cancer incidence and mortality. Breast Cancer Res. 2004;6(6):229-39. doi: 10.1186/bcr932. Epub 2004 Aug 26. PMID 15535852
- [Background] Brunt AM, Wheatley D, Yarnold J, Somaiah N, Kelly S, Harnett A, Coles C, Goodman A, Bahl A, Churn M, Zotova R, Sydenham M, Griffin CL, Morden JP, Bliss JM; FAST-Forward Trial Management Group. Acute skin toxicity associated with a 1-week schedule of whole breast radiotherapy compared with a standard 3-week regimen delivered in the UK FAST-Forward Trial. Radiother Oncol. 2016 Jul;120(1):114-8. doi: 10.1016/j.radonc.2016.02.027. Epub 2016 Apr 1. PMID 27046390
- [Background] Brunt AM, Haviland JS, Sydenham M, Agrawal RK, Algurafi H, Alhasso A, Barrett-Lee P, Bliss P, Bloomfield D, Bowen J, Donovan E, Goodman A, Harnett A, Hogg M, Kumar S, Passant H, Quigley M, Sherwin L, Stewart A, Syndikus I, Tremlett J, Tsang Y, Venables K, Wheatley D, Bliss JM, Yarnold JR. Ten-Year Results of FAST: A Randomized Controlled Trial of 5-Fraction Whole-Breast Radiotherapy for Early Breast Cancer. J Clin Oncol. 2020 Oct 1;38(28):3261-3272. doi: 10.1200/JCO.19.02750. Epub 2020 Jul 14. PMID 32663119
- [Background] Chan EK, Woods R, Virani S, Speers C, Wai ES, Nichol A, McBride ML, Tyldesley S. Long-term mortality from cardiac causes after adjuvant hypofractionated vs. conventional radiotherapy for localized left-sided breast cancer. Radiother Oncol. 2015 Jan;114(1):73-8. doi: 10.1016/j.radonc.2014.08.021. Epub 2014 Sep 13. PMID 25227961
- [Background] Perou CM, Sorlie T, Eisen MB, van de Rijn M, Jeffrey SS, Rees CA, Pollack JR, Ross DT, Johnsen H, Akslen LA, Fluge O, Pergamenschikov A, Williams C, Zhu SX, Lonning PE, Borresen-Dale AL, Brown PO, Botstein D. Molecular portraits of human breast tumours. Nature. 2000 Aug 17;406(6797):747-52. doi: 10.1038/35021093. PMID 10963602
- [Background] Ciammella P, Podgornii A, Galeandro M, Micera R, Ramundo D, Palmieri T, Cagni E, Iotti C. Toxicity and cosmetic outcome of hypofractionated whole-breast radiotherapy: predictive clinical and dosimetric factors. Radiat Oncol. 2014 Apr 24;9:97. doi: 10.1186/1748-717X-9-97. PMID 24762173
- [Background] Clavel-Chapelon F, Gerber M. Reproductive factors and breast cancer risk. Do they differ according to age at diagnosis? Breast Cancer Res Treat. 2002 Mar;72(2):107-15. doi: 10.1023/a:1014891216621. PMID 12038701
- [Background] Cox JD, Stetz J, Pajak TF. Toxicity criteria of the Radiation Therapy Oncology Group (RTOG) and the European Organization for Research and Treatment of Cancer (EORTC). Int J Radiat Oncol Biol Phys. 1995 Mar 30;31(5):1341-6. doi: 10.1016/0360-3016(95)00060-C. No abstract available. PMID 7713792
- [Background] Early Breast Cancer Trialists' Collaborative Group (EBCTCG); Darby S, McGale P, Correa C, Taylor C, Arriagada R, Clarke M, Cutter D, Davies C, Ewertz M, Godwin J, Gray R, Pierce L, Whelan T, Wang Y, Peto R. Effect of radiotherapy after breast-conserving surgery on 10-year recurrence and 15-year breast cancer death: meta-analysis of individual patient data for 10,801 women in 17 randomised trials. Lancet. 2011 Nov 12;378(9804):1707-16. doi: 10.1016/S0140-6736(11)61629-2. Epub 2011 Oct 19. PMID 22019144
- [Background] Early Breast Cancer Trialists' Collaborative Group. Effects of radiotherapy and surgery in early breast cancer. An overview of the randomized trials. N Engl J Med. 1995 Nov 30;333(22):1444-55. doi: 10.1056/NEJM199511303332202. PMID 7477144
- [Background] Fiolet T, Srour B, Sellem L, Kesse-Guyot E, Alles B, Mejean C, Deschasaux M, Fassier P, Latino-Martel P, Beslay M, Hercberg S, Lavalette C, Monteiro CA, Julia C, Touvier M. Consumption of ultra-processed foods and cancer risk: results from NutriNet-Sante prospective cohort. BMJ. 2018 Feb 14;360:k322. doi: 10.1136/bmj.k322. PMID 29444771
- [Background] Fisher B, Anderson S, Bryant J, Margolese RG, Deutsch M, Fisher ER, Jeong JH, Wolmark N. Twenty-year follow-up of a randomized trial comparing total mastectomy, lumpectomy, and lumpectomy plus irradiation for the treatment of invasive breast cancer. N Engl J Med. 2002 Oct 17;347(16):1233-41. doi: 10.1056/NEJMoa022152. PMID 12393820
- [Background] Folkerd E, Dowsett M. Sex hormones and breast cancer risk and prognosis. Breast. 2013 Aug;22 Suppl 2:S38-43. doi: 10.1016/j.breast.2013.07.007. PMID 24074790
- [Background] Fragomeni SM, Sciallis A, Jeruss JS. Molecular Subtypes and Local-Regional Control of Breast Cancer. Surg Oncol Clin N Am. 2018 Jan;27(1):95-120. doi: 10.1016/j.soc.2017.08.005. PMID 29132568
- [Background] Grann VR, Panageas KS, Whang W, Antman KH, Neugut AI. Decision analysis of prophylactic mastectomy and oophorectomy in BRCA1-positive or BRCA2-positive patients. J Clin Oncol. 1998 Mar;16(3):979-85. doi: 10.1200/JCO.1998.16.3.979. PMID 9508180
- [Background] HALL, E. J. .; GIACCIA, A. J. Radiobiology for the Radiologist - Eighth Edition. [s.l.] Wolters Kluwer, 2019. v. 148
- [Background] HALPERIN, E. C. et al. Perez & Brady's Principles and Practice of Radiation Oncology, Sixth Edition- Halperin, Edward C,. 6th. ed. [s.l: s.n.].
- [Background] Hancke K, Denkinger MD, Konig J, Kurzeder C, Wockel A, Herr D, Blettner M, Kreienberg R. Standard treatment of female patients with breast cancer decreases substantially for women aged 70 years and older: a German clinical cohort study. Ann Oncol. 2010 Apr;21(4):748-753. doi: 10.1093/annonc/mdp364. Epub 2009 Oct 13. PMID 19825884
- [Background] Haviland JS, Owen JR, Dewar JA, Agrawal RK, Barrett J, Barrett-Lee PJ, Dobbs HJ, Hopwood P, Lawton PA, Magee BJ, Mills J, Simmons S, Sydenham MA, Venables K, Bliss JM, Yarnold JR; START Trialists' Group. The UK Standardisation of Breast Radiotherapy (START) trials of radiotherapy hypofractionation for treatment of early breast cancer: 10-year follow-up results of two randomised controlled trials. Lancet Oncol. 2013 Oct;14(11):1086-1094. doi: 10.1016/S1470-2045(13)70386-3. Epub 2013 Sep 19. PMID 24055415
- [Background] Hickey BE, James ML, Lehman M, Hider PN, Jeffery M, Francis DP, See AM. Fraction size in radiation therapy for breast conservation in early breast cancer. Cochrane Database Syst Rev. 2016 Jul 18;7(7):CD003860. doi: 10.1002/14651858.CD003860.pub4. PMID 27425588
- [Background] Hill DA, Prossnitz ER, Royce M, Nibbe A. Temporal trends in breast cancer survival by race and ethnicity: A population-based cohort study. PLoS One. 2019 Oct 24;14(10):e0224064. doi: 10.1371/journal.pone.0224064. eCollection 2019. PMID 31647839
- [Background] Hoffman-Goetz L, Apter D, Demark-Wahnefried W, Goran MI, McTiernan A, Reichman ME. Possible mechanisms mediating an association between physical activity and breast cancer. Cancer. 1998 Aug 1;83(3 Suppl):621-8. doi: 10.1002/(sici)1097-0142(19980801)83:3+3.0.co;2-a. PMID 9690525
- [Background] INSTITUTO NACIONAL DE CÂNCER; JOSÉ ALENCAR GOMES DA SILVA. Estimativa 2020: incidência de câncer no Brasil. [s.l: s.n.].
- [Background] Kolb R, Zhang W. Obesity and Breast Cancer: A Case of Inflamed Adipose Tissue. Cancers (Basel). 2020 Jun 25;12(6):1686. doi: 10.3390/cancers12061686. PMID 32630445
- [Background] Lalani N, Voduc KD, Jimenez RB, Levasseur N, Gondara L, Speers C, Lohrisch C, Nichol A. Breast Cancer Molecular Subtype as a Predictor of Radiation Therapy Fractionation Sensitivity. Int J Radiat Oncol Biol Phys. 2021 Jan 1;109(1):281-287. doi: 10.1016/j.ijrobp.2020.08.038. Epub 2020 Aug 24. PMID 32853707
- [Background] Lowery AJ, Kell MR, Glynn RW, Kerin MJ, Sweeney KJ. Locoregional recurrence after breast cancer surgery: a systematic review by receptor phenotype. Breast Cancer Res Treat. 2012 Jun;133(3):831-41. doi: 10.1007/s10549-011-1891-6. Epub 2011 Dec 7. PMID 22147079
- [Background] Lukasiewicz S, Czeczelewski M, Forma A, Baj J, Sitarz R, Stanislawek A. Breast Cancer-Epidemiology, Risk Factors, Classification, Prognostic Markers, and Current Treatment Strategies-An Updated Review. Cancers (Basel). 2021 Aug 25;13(17):4287. doi: 10.3390/cancers13174287. PMID 34503097
- [Background] Lux MP, Fasching PA, Beckmann MW. Hereditary breast and ovarian cancer: review and future perspectives. J Mol Med (Berl). 2006 Jan;84(1):16-28. doi: 10.1007/s00109-005-0696-7. Epub 2005 Nov 11. PMID 16283147
- [Background] Macacu A, Autier P, Boniol M, Boyle P. Active and passive smoking and risk of breast cancer: a meta-analysis. Breast Cancer Res Treat. 2015 Nov;154(2):213-24. doi: 10.1007/s10549-015-3628-4. Epub 2015 Nov 6. PMID 26546245
- [Background] MACDONALD, S. et al. Breast Contouring RADCOMP Consortium, 2016. Disponível em: <https://www.rtog.org/corelab/contouringatlases.aspx>
- [Background] Marta GN, Coles C, Kaidar-Person O, Meattini I, Hijal T, Zissiadis Y, Pignol JP, Ramiah D, Ho AY, Cheng SH, Sancho G, Offersen BV, Poortmans P. The use of moderately hypofractionated post-operative radiation therapy for breast cancer in clinical practice: A critical review. Crit Rev Oncol Hematol. 2020 Dec;156:103090. doi: 10.1016/j.critrevonc.2020.103090. Epub 2020 Aug 26. PMID 33091800
- [Background] Marta GN, Riera R, Pacheco RL, Cabrera Martimbianco AL, Meattini I, Kaidar-Person O, Poortmans P. Moderately hypofractionated post-operative radiation therapy for breast cancer: Systematic review and meta-analysis of randomized clinical trials. Breast. 2022 Apr;62:84-92. doi: 10.1016/j.breast.2022.01.018. Epub 2022 Feb 3. PMID 35131647
- [Background] EBCTCG (Early Breast Cancer Trialists' Collaborative Group); McGale P, Taylor C, Correa C, Cutter D, Duane F, Ewertz M, Gray R, Mannu G, Peto R, Whelan T, Wang Y, Wang Z, Darby S. Effect of radiotherapy after mastectomy and axillary surgery on 10-year recurrence and 20-year breast cancer mortality: meta-analysis of individual patient data for 8135 women in 22 randomised trials. Lancet. 2014 Jun 21;383(9935):2127-35. doi: 10.1016/S0140-6736(14)60488-8. Epub 2014 Mar 19. PMID 24656685
- [Background] Meattini I, Becherini C, Boersma L, Kaidar-Person O, Marta GN, Montero A, Offersen BV, Aznar MC, Belka C, Brunt AM, Dicuonzo S, Franco P, Krause M, MacKenzie M, Marinko T, Marrazzo L, Ratosa I, Scholten A, Senkus E, Stobart H, Poortmans P, Coles CE. European Society for Radiotherapy and Oncology Advisory Committee in Radiation Oncology Practice consensus recommendations on patient selection and dose and fractionation for external beam radiotherapy in early breast cancer. Lancet Oncol. 2022 Jan;23(1):e21-e31. doi: 10.1016/S1470-2045(21)00539-8. PMID 34973228
- [Background] Mendez LC, Moraes FY, Fernandes GDS, Weltman E. Cancer Deaths due to Lack of Universal Access to Radiotherapy in the Brazilian Public Health System. Clin Oncol (R Coll Radiol). 2018 Jan;30(1):e29-e36. doi: 10.1016/j.clon.2017.09.003. Epub 2017 Oct 5. PMID 28988891
- [Background] Monten C, Lievens Y, Olteanu LAM, Paelinck L, Speleers B, Deseyne P, Van Den Broecke R, De Neve W, Veldeman L. Highly Accelerated Irradiation in 5 Fractions (HAI-5): Feasibility in Elderly Women With Early or Locally Advanced Breast Cancer. Int J Radiat Oncol Biol Phys. 2017 Jul 15;98(4):922-930. doi: 10.1016/j.ijrobp.2017.01.229. Epub 2017 Feb 1. PMID 28366576
- [Background] Moraes FY, Marta GN, Hanna SA, Leite ET, Ferrigno R, da Silva JL, Carvalho Hde A. Brazil's Challenges and Opportunities. Int J Radiat Oncol Biol Phys. 2015 Jul 15;92(4):707-12. doi: 10.1016/j.ijrobp.2014.12.063. No abstract available. PMID 26104923
- [Background] Morrow M, Strom EA, Bassett LW, Dershaw DD, Fowble B, Harris Ja, O'Malley F, Schnitt SJ, Singletary SE, Winchester DP; American College of Surgeons; College of American Pathology; Society of Surgical Oncology; American College of Radiology. Standard for the management of ductal carcinoma in situ of the breast (DCIS). CA Cancer J Clin. 2002 Sep-Oct;52(5):256-76. doi: 10.3322/canjclin.52.5.256. PMID 12363325
- [Background] Murray Brunt A, Haviland JS, Wheatley DA, Sydenham MA, Alhasso A, Bloomfield DJ, Chan C, Churn M, Cleator S, Coles CE, Goodman A, Harnett A, Hopwood P, Kirby AM, Kirwan CC, Morris C, Nabi Z, Sawyer E, Somaiah N, Stones L, Syndikus I, Bliss JM, Yarnold JR; FAST-Forward Trial Management Group. Hypofractionated breast radiotherapy for 1 week versus 3 weeks (FAST-Forward): 5-year efficacy and late normal tissue effects results from a multicentre, non-inferiority, randomised, phase 3 trial. Lancet. 2020 May 23;395(10237):1613-1626. doi: 10.1016/S0140-6736(20)30932-6. Epub 2020 Apr 28. PMID 32580883
- [Background] Narod SA. Hormone replacement therapy and the risk of breast cancer. Nat Rev Clin Oncol. 2011 Aug 2;8(11):669-76. doi: 10.1038/nrclinonc.2011.110. PMID 21808267
- [Background] Offersen BV, Alsner J, Nielsen HM, Jakobsen EH, Nielsen MH, Krause M, Stenbygaard L, Mjaaland I, Schreiber A, Kasti UM, Overgaard J; Danish Breast Cancer Group Radiation Therapy Committee. Hypofractionated Versus Standard Fractionated Radiotherapy in Patients With Early Breast Cancer or Ductal Carcinoma In Situ in a Randomized Phase III Trial: The DBCG HYPO Trial. J Clin Oncol. 2020 Nov 1;38(31):3615-3625. doi: 10.1200/JCO.20.01363. Epub 2020 Sep 10. PMID 32910709
- [Background] Ortholan C, Hannoun-Levi JM, Ferrero JM, Largillier R, Courdi A. Long-term results of adjuvant hypofractionated radiotherapy for breast cancer in elderly patients. Int J Radiat Oncol Biol Phys. 2005 Jan 1;61(1):154-62. doi: 10.1016/j.ijrobp.2004.04.059. PMID 15629606
- [Background] Owen JR, Ashton A, Bliss JM, Homewood J, Harper C, Hanson J, Haviland J, Bentzen SM, Yarnold JR. Effect of radiotherapy fraction size on tumour control in patients with early-stage breast cancer after local tumour excision: long-term results of a randomised trial. Lancet Oncol. 2006 Jun;7(6):467-71. doi: 10.1016/S1470-2045(06)70699-4. PMID 16750496
- [Background] Porter P. "Westernizing" women's risks? Breast cancer in lower-income countries. N Engl J Med. 2008 Jan 17;358(3):213-6. doi: 10.1056/NEJMp0708307. No abstract available. PMID 18199859
- [Background] Recht A, Comen EA, Fine RE, Fleming GF, Hardenbergh PH, Ho AY, Hudis CA, Hwang ES, Kirshner JJ, Morrow M, Salerno KE, Sledge GW Jr, Solin LJ, Spears PA, Whelan TJ, Somerfield MR, Edge SB. Postmastectomy Radiotherapy: An American Society of Clinical Oncology, American Society for Radiation Oncology, and Society of Surgical Oncology Focused Guideline Update. J Clin Oncol. 2016 Dec 20;34(36):4431-4442. doi: 10.1200/JCO.2016.69.1188. Epub 2016 Sep 30. PMID 27646947
- [Background] Salmon RJ, Remvikos Y, Campana F, Languille O, Magdalenat H, Asselain B, Clough KB; Breast Group of the Institut Curie. Neo adjuvant Tamoxifen in post menopausal patients with operable breast cancer. Eur J Surg Oncol. 2003 Dec;29(10):831-4. doi: 10.1016/s0748-7983(03)00095-7. PMID 14624772
- [Background] Sharma R. Breast cancer incidence, mortality and mortality-to-incidence ratio (MIR) are associated with human development, 1990-2016: evidence from Global Burden of Disease Study 2016. Breast Cancer. 2019 Jul;26(4):428-445. doi: 10.1007/s12282-018-00941-4. Epub 2019 Jan 2. PMID 30604398
- [Background] Siegel R, Ma J, Zou Z, Jemal A. Cancer statistics, 2014. CA Cancer J Clin. 2014 Jan-Feb;64(1):9-29. doi: 10.3322/caac.21208. Epub 2014 Jan 7. PMID 24399786
- [Background] Smith BD, Bellon JR, Blitzblau R, Freedman G, Haffty B, Hahn C, Halberg F, Hoffman K, Horst K, Moran J, Patton C, Perlmutter J, Warren L, Whelan T, Wright JL, Jagsi R. Radiation therapy for the whole breast: Executive summary of an American Society for Radiation Oncology (ASTRO) evidence-based guideline. Pract Radiat Oncol. 2018 May-Jun;8(3):145-152. doi: 10.1016/j.prro.2018.01.012. Epub 2018 Mar 12. PMID 29545124
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Swerdlow AJ, Cooke R, Bates A, Cunningham D, Falk SJ, Gilson D, Hancock BW, Harris SJ, Horwich A, Hoskin PJ, Linch DC, Lister TA, Lucraft HH, Radford JA, Stevens AM, Syndikus I, Williams MV. Breast cancer risk after supradiaphragmatic radiotherapy for Hodgkin's lymphoma in England and Wales: a National Cohort Study. J Clin Oncol. 2012 Aug 1;30(22):2745-52. doi: 10.1200/JCO.2011.38.8835. Epub 2012 Jun 25. PMID 22734026
- [Background] Taylor P, Castilho MS, Marta GN. Cost containment analysis and access to treatment associated with adopting hypofractionated radiation therapy from the Brazilian perspective. Lancet Reg Health Am. 2022 Jun 9;13:100292. doi: 10.1016/j.lana.2022.100292. eCollection 2022 Sep. PMID 36777322
- [Background] START Trialists' Group; Bentzen SM, Agrawal RK, Aird EG, Barrett JM, Barrett-Lee PJ, Bliss JM, Brown J, Dewar JA, Dobbs HJ, Haviland JS, Hoskin PJ, Hopwood P, Lawton PA, Magee BJ, Mills J, Morgan DA, Owen JR, Simmons S, Sumo G, Sydenham MA, Venables K, Yarnold JR. The UK Standardisation of Breast Radiotherapy (START) Trial A of radiotherapy hypofractionation for treatment of early breast cancer: a randomised trial. Lancet Oncol. 2008 Apr;9(4):331-41. doi: 10.1016/S1470-2045(08)70077-9. Epub 2008 Mar 19. PMID 18356109
- [Background] Trombetta M, Julian TB, Werts ED, Colonias A, Betler J, Kotinsley K, Kim Y, Parda D. Comparison of conservative management techniques in the re-treatment of ipsilateral breast tumor recurrence. Brachytherapy. 2011 Jan-Feb;10(1):74-80. doi: 10.1016/j.brachy.2010.01.005. Epub 2010 Aug 4. PMID 20685174
- [Background] U.S. DEPARTMENT OF HEALTH AND HUMAN SERVICES. Common Terminology Criteria for Adverse Events (CTCAE).v.5.0. Cancer Therapy Evaluation Program (CTEP), 2017.
- [Background] Truong PT, Bernstein V, Lesperance M, Speers CH, Olivotto IA. Radiotherapy omission after breast-conserving surgery is associated with reduced breast cancer-specific survival in elderly women with breast cancer. Am J Surg. 2006 Jun;191(6):749-55. doi: 10.1016/j.amjsurg.2005.07.028. PMID 16720143
- [Background] Verbanck S, Hanon S, Schuermans D, Van Parijs H, Vinh-Hung V, Miedema G, Verellen D, Storme G, Fontaine C, Lamote J, De Ridder M, Vincken W. Mild Lung Restriction in Breast Cancer Patients After Hypofractionated and Conventional Radiation Therapy: A 3-Year Follow-Up. Int J Radiat Oncol Biol Phys. 2016 Jul 1;95(3):937-945. doi: 10.1016/j.ijrobp.2016.02.008. Epub 2016 Feb 6. PMID 27302510
- [Background] Veronesi U, Cascinelli N, Mariani L, Greco M, Saccozzi R, Luini A, Aguilar M, Marubini E. Twenty-year follow-up of a randomized study comparing breast-conserving surgery with radical mastectomy for early breast cancer. N Engl J Med. 2002 Oct 17;347(16):1227-32. doi: 10.1056/NEJMoa020989. PMID 12393819
- [Background] Visvader JE, Stingl J. Mammary stem cells and the differentiation hierarchy: current status and perspectives. Genes Dev. 2014 Jun 1;28(11):1143-58. doi: 10.1101/gad.242511.114. PMID 24888586
- [Background] Visvanathan K, Hurley P, Bantug E, Brown P, Col NF, Cuzick J, Davidson NE, Decensi A, Fabian C, Ford L, Garber J, Katapodi M, Kramer B, Morrow M, Parker B, Runowicz C, Vogel VG 3rd, Wade JL, Lippman SM. Use of pharmacologic interventions for breast cancer risk reduction: American Society of Clinical Oncology clinical practice guideline. J Clin Oncol. 2013 Aug 10;31(23):2942-62. doi: 10.1200/JCO.2013.49.3122. Epub 2013 Jul 8. PMID 23835710
- [Background] Visvanathan K, Fabian CJ, Bantug E, Brewster AM, Davidson NE, DeCensi A, Floyd JD, Garber JE, Hofstatter EW, Khan SA, Katapodi MC, Pruthi S, Raab R, Runowicz CD, Somerfield MR. Use of Endocrine Therapy for Breast Cancer Risk Reduction: ASCO Clinical Practice Guideline Update. J Clin Oncol. 2019 Nov 20;37(33):3152-3165. doi: 10.1200/JCO.19.01472. Epub 2019 Sep 3. PMID 31479306
- [Background] Vrieling C, van Werkhoven E, Maingon P, Poortmans P, Weltens C, Fourquet A, Schinagl D, Oei B, Rodenhuis CC, Horiot JC, Struikmans H, Van Limbergen E, Kirova Y, Elkhuizen P, Bongartz R, Miralbell R, Morgan DA, Dubois JB, Remouchamps V, Mirimanoff RO, Hart G, Collette S, Collette L, Bartelink H; European Organisation for Research and Treatment of Cancer, Radiation Oncology and Breast Cancer Groups. Prognostic Factors for Local Control in Breast Cancer After Long-term Follow-up in the EORTC Boost vs No Boost Trial: A Randomized Clinical Trial. JAMA Oncol. 2017 Jan 1;3(1):42-48. doi: 10.1001/jamaoncol.2016.3031. PMID 27607734
- [Background] Waks AG, Winer EP. Breast Cancer Treatment: A Review. JAMA. 2019 Jan 22;321(3):288-300. doi: 10.1001/jama.2018.19323. PMID 30667505
- [Background] Wang SL, Fang H, Song YW, Wang WH, Hu C, Liu YP, Jin J, Liu XF, Yu ZH, Ren H, Li N, Lu NN, Tang Y, Tang Y, Qi SN, Sun GY, Peng R, Li S, Chen B, Yang Y, Li YX. Hypofractionated versus conventional fractionated postmastectomy radiotherapy for patients with high-risk breast cancer: a randomised, non-inferiority, open-label, phase 3 trial. Lancet Oncol. 2019 Mar;20(3):352-360. doi: 10.1016/S1470-2045(18)30813-1. Epub 2019 Jan 30. PMID 30711522
- [Background] Wang SL, Fang H, Hu C, Song YW, Wang WH, Jin J, Liu YP, Ren H, Liu J, Li GF, Du XH, Tang Y, Jing H, Ma YC, Huang Z, Chen B, Tang Y, Li N, Lu NN, Qi SN, Yang Y, Sun GY, Liu XF, Li YX. Hypofractionated Versus Conventional Fractionated Radiotherapy After Breast-Conserving Surgery in the Modern Treatment Era: A Multicenter, Randomized Controlled Trial From China. J Clin Oncol. 2020 Nov 1;38(31):3604-3614. doi: 10.1200/JCO.20.01024. Epub 2020 Aug 11. PMID 32780661
- [Background] Weiss A, Noorbakhsh A, Tokin C, Chang D, Blair SL. Hormone receptor-negative breast cancer: undertreatment of patients over 80. Ann Surg Oncol. 2013 Oct;20(10):3274-8. doi: 10.1245/s10434-013-3115-2. Epub 2013 Jul 10. PMID 23838924
- [Background] Weltman E, Marta GN. Radiotherapy and the SUS: A collapse foretold. Rev Assoc Med Bras (1992). 2017 Feb;63(2):93-94. doi: 10.1590/1806-9282.63.02.93. No abstract available. PMID 28355367
- [Background] Whelan T, MacKenzie R, Julian J, Levine M, Shelley W, Grimard L, Lada B, Lukka H, Perera F, Fyles A, Laukkanen E, Gulavita S, Benk V, Szechtman B. Randomized trial of breast irradiation schedules after lumpectomy for women with lymph node-negative breast cancer. J Natl Cancer Inst. 2002 Aug 7;94(15):1143-50. doi: 10.1093/jnci/94.15.1143. PMID 12165639
- [Background] Whelan TJ, Pignol JP, Levine MN, Julian JA, MacKenzie R, Parpia S, Shelley W, Grimard L, Bowen J, Lukka H, Perera F, Fyles A, Schneider K, Gulavita S, Freeman C. Long-term results of hypofractionated radiation therapy for breast cancer. N Engl J Med. 2010 Feb 11;362(6):513-20. doi: 10.1056/NEJMoa0906260. PMID 20147717
- [Background] Winters S, Martin C, Murphy D, Shokar NK. Breast Cancer Epidemiology, Prevention, and Screening. Prog Mol Biol Transl Sci. 2017;151:1-32. doi: 10.1016/bs.pmbts.2017.07.002. Epub 2017 Oct 10. PMID 29096890
- [Background] WHO Position Paper on Mammography Screening. Geneva: World Health Organization; 2014. Available from http://www.ncbi.nlm.nih.gov/books/NBK269545/ PMID 25642524
- [Background] Yarnold J, Ashton A, Bliss J, Homewood J, Harper C, Hanson J, Haviland J, Bentzen S, Owen R. Fractionation sensitivity and dose response of late adverse effects in the breast after radiotherapy for early breast cancer: long-term results of a randomised trial. Radiother Oncol. 2005 Apr;75(1):9-17. doi: 10.1016/j.radonc.2005.01.005. Epub 2005 Mar 16. PMID 15878095
- [Background] FAST Trialists group; Agrawal RK, Alhasso A, Barrett-Lee PJ, Bliss JM, Bliss P, Bloomfield D, Bowen J, Brunt AM, Donovan E, Emson M, Goodman A, Harnett A, Haviland JS, Kaggwa R, Morden JP, Robinson A, Simmons S, Stewart A, Sydenham MA, Syndikus I, Tremlett J, Tsang Y, Wheatley D, Venables K, Yarnold JR. First results of the randomised UK FAST Trial of radiotherapy hypofractionation for treatment of early breast cancer (CRUKE/04/015). Radiother Oncol. 2011 Jul;100(1):93-100. doi: 10.1016/j.radonc.2011.06.026. PMID 21752481
- [Derived] Fang M, Gico VC, Casimiro L, Takatsu B, Santos Neto E, Mendoza Lopez RV, Costa Pinto GV, Marta GN. Phase II Evaluation of Ultra-Hypofractionated Postoperative Radiation Therapy for Breast Cancer: Toxicity and Efficacy in a Single-Center Nonrandomized Prospective Study. JCO Glob Oncol. 2025 Mar;11:e2400277. doi: 10.1200/GO-24-00277. Epub 2025 Mar 7. PMID 40053900